CLINICAL TRIAL: NCT06253611
Title: Gut Microbiome Intervention With EXL01 in Combination With Nivolumab and FOLFOX as First-line Treatment for Patients With PD-L1 CPS ≥5 Metastatic Gastric Cancer: A Randomized GERCOR Phase II Study (BIG)
Brief Title: First-line EXL01 With Nivolumab and FOLFOX for PD-L1 CPS ≥5 Metastatic Gastric Cancer
Acronym: BIG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIG G-122 PRODIGE 94
Record Dates: First submitted 2024-01-31; First posted 2024-02-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; Folfox protocol; Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab Combined With FOLFOX and EXL01 (Experimental): Nivolumab 240 mg IV q2w and FOLFOX q2w plus EXL01 orally once daily
  Interventions: Drug: Nivolumab; Drug: FOLFOX regimen; Biological: EXL01
- Nivolumab and FOLFOX (Active Comparator): Nivolumab 240 mg IV q2w and FOLFOX q2w
  Interventions: Drug: Nivolumab; Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240 mg IV; every 2 weeks
  Other Names: Opdivo
Drug: FOLFOX regimen — Oxaliplatin 85 mg/m², leucovorin 400 mg/m², bolus of 5-FU 400 mg/m², continuous 5-FU 2400/m² in 46 hours; every 2 weeks
  Other Names: Leucovorin, fluorouracil, and oxaliplatin
Biological: EXL01 — Orally 1 capsule/day, starting on day 1 of each FOLFOX/nivolumab treatment.
  Arms: Nivolumab Combined With FOLFOX and EXL01

SUMMARY:
This is a randomized non-comparative, multicenter phase II study in patients with PD-L1 PD-L1 combined positive score (CPS) ≥5 advanced gastric cancer to evaluate the efficacy and safety of nivolumab and FOLFOX in combination with EXL01 as first-line treatment.

After signing the informed consent form, and upon confirmation of the patient's eligibility, patients will be randomized in a 2:1 ratio to either the nivolumab and FOLFOX plus EXL01 arm (experimental) or the nivolumab and FOLFOX arm (control). In both arms, treatment will be given until PD, unacceptable toxicity or for a maximum of 24 months (52 cycles).

DETAILED DESCRIPTION:
The primary objective of the study is to assess the objective response rate (ORR) at 4 months (based on Response Evaluation Criteria in Solid Tumor [RECIST] criteria v1.1) of patients with PD-L1 CPS ≥ 5 advanced gastric cancer treated by EXL01 plus nivolumab and FOLFOX as first-line treatment.

With a randomization ratio of 2:1 it will be necessary to randomize 40 patients in the control arm, 80 patients in the experimental arm and so a total of 120 evaluable patients in the study. Randomization will be stratified by PD-L1 expression level, center, and prior gastrectomy.

In the experimental arm, the primary analysis will be on modified intent-to-treat (mITT) population. Confirmative analysis will be conducted firstly in the ITT population and secondly, in the Per Protocol (PP). Analyses of safety will be conducted in safety population.

The Kaplan-Meier method will be used to estimate time to event endpoints and described using the median and event-free rates over time with CI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have dated and signed an approved written informed consent form. This must be obtained before the performance of any protocol-related procedures that are not part of normal patient care.
2. Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study,

   Target Population
3. Inoperable, advanced, or metastatic gastric cancer or gastroesophageal junction or distal esophageal carcinoma and histologically confirmed predominant adenocarcinoma,
4. Expression of PD-L1 with a combined positive score (PD-L1 CPS) ≥5, Note: information must be available at the time of inclusion, the examination will be performed locally in the center and secondarily confirmed centrally,
5. No prior systemic cancer treatment given as primary therapy for advanced nonresectable or metastatic disease, Note: if patient received neoadjuvant/adjuvant therapy, this therapy should be completed at least 6 months prior to the diagnosis of metastatic or recurrent disease is made. Palliative radiotherapy is allowed and must be completed 2 weeks prior to randomization,
6. At least one measurable lesion as assessed by computed tomography (CT)-scan or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and feasibility of repeated radiological assessments; radiographic tumor assessment should be performed within 28 days prior to randomization,
7. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1,
8. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to randomization of study treatment:

   1. White blood cell ≥ 2000/μL;
   2. Neutrophils ≥ 2000/μL;
   3. Platelets ≥ 100.000/μL;
   4. Hemoglobin ≥ 9.0 g/dL;
   5. Serum albumin ≥ 30 g/L;
   6. Serum creatinine level ≤ 150 μM and calculated creatinine clearance (Cockcroft-Gault) > 50 mL/minute,
   7. Total bilirubin ≤ 1.5 x upper normal limit (ULN);
   8. Alanine aminotransferase (ALT) ≤ 3.0 x ULN (or ≤ 5.0 x ULN if liver metastases are present);
   9. Aspartame aminotransferase (AST) ≤ 3.0 x ULN (or ≤ 5.0 x ULN if liver metastases are present);
   10. Potassium ≥ 1.0 x lower limit of normal (LLN),
   11. Magnesium ≥ 1.0 x LLN,
   12. Calcium ≥ 1.0 x LLN,
9. Baseline-corrected QT interval ≤ 450 msec for males and ≤ 470 msec for females,
10. Availability of a representative tumor tissue specimen for exploratory translational research; tumor tissue samples, either formalin- fixed paraffin-embedded (FFPE) tissue block or unstained tumor tissue sections (minimum of 20 positively charged slides) from primary or metastatic site must be submitted to the central laboratory,
11. Registration in a national health care system (PUMa-Protection Universelle Maladie included.

    Age and reproductive status
12. Age ≥ 18 years,
13. Women must not be pregnant, breastfeeding, or expecting to conceive during the study,
14. Reproductive status:

    1. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the start of study drug,
    2. WOCBP must agree to use an adequate method of contraception or birth control for the duration of study treatment and 5 months (nivolumab), 9 months (oxaliplatin), 6 months (5-FU) or at least 1 month (EXL01) of the patient's last dose of the study drug,
    3. Males who are fertile and sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment and 6 months (nivolumab, oxaliplatin, or 5-FU) or at least 1 month (EXL01) after the last dose of study treatment. In addition, males must be willing to refrain from sperm donation during this time,

Exclusion Criteria:

Target Disease Exceptions

1. Known HER-2 positive status or unknown HER-2 status before inclusion,
2. Active brain metastases or known history of leptomeningeal carcinomatosis,
3. Ascites, which cannot be controlled with appropriate interventions,

   Exclusion criteria related to medical history and concurrent disease
4. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast,
5. Active, known, or suspected autoimmune disease; type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted,
6. Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity,
7. Prior treatment with an anti-PD(L)1, anti-LAG-3, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co- stimulation or immune checkpoint pathways, including prior therapy with anti-tumor vaccines or other immuno-stimulatory antitumor agents,
8. Condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days (2 weeks) of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, are permitted prior to randomization in the absence of active autoimmune disease,
9. Persistence of toxicity (The National Cancer Institute Common Terminology Criteria for Adverse Event [NCI CTCAE] v 5.0) grade >1 related to prior anticancer treatments,
10. Major surgery within 28 days (4 weeks) prior to first dose of study treatment, Note: Participants who had surgery >4 weeks prior to screening must have recovered adequately from any toxicity and/or complications from the surgery or trauma prior to starting study intervention.
11. Concomitant unplanned antitumor therapy (e.g., chemotherapy, molecular targeted therapy, radiotherapy, immunotherapy),

    Exclusion criteria related to EXL01
12. GI obstruction, poor oral intake, or difficulty in taking oral medication or difficulties in swallowing; nasogastric tubes are not permitted,
13. Known GI malabsorption,
14. Is currently participating in or has participated in a study with an investigational compound within 28 days prior to the first dose of study treatment, Note: Participants who have entered the follow-up phase of an investigational study may participate so long as it has been at least 3 months since the last dose of the previous investigational agent,
15. Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
16. Fecal microbiota transplant within 3 months prior to screening, Note: Patients must have recovered adequately from the toxicity and/or complications from the treatment prior to starting study intervention.
17. Current probiotics administration, or planned probiotics administration during treatment course is not allowed, Note: The following therapies should be avoided during the study; however, they are not prohibited if, in the assessment of the

    Investigator, they are required for clinical management:
    * Nonsteroidal anti-inflammatories,
    * Antacids,
    * Proton-pump inhibitors.
18. Excessive alcohol intake: moderate consumption, defined as no more than 1 drink per day for women and no more than 2 drinks per day for men, is permitted,
19. Known allergy and/or hypersensitivity to any component or excipients of study treatments (nivolumab, EXL01), any other live pro- biotherapeutic product, and/or to soybean or soy-containing products,
20. Known history or newly diagnosed GI parasitic infection within 3 months prior to screening, Note: Patients must have recovered adequately from the toxicity and/or complications from the treatment prior to starting study intervention,
21. Active inflammatory intestinal disease (Crohn disease, Hemorrhagic recto-colitis, coeliac disease) or any serious chronic intestinal disease with uncontrolled diarrhea, or other inflammatory disease requiring anti-inflammatory medications (according to exclusion criteria n°8),

    Exclusion criteria related to chemotherapy
22. Active or chronic hepatitis B virus (HBV), hepatitis C virus (HCV) and/or human immunodeficiency virus infection (HIV 1/2 antibodies).

    Participants are eligible if they:
    * Have controlled HCV load defined as undetectable hepatitis C RNA by polymerase chain reaction either spontaneously or in response to a successful prior course of anti-hepatitis C therapy,
    * Have received HBV vaccination with only anti-HBs positivity and no clinical signs of hepatitis,
    * Are HBV surface antigen (HBsAg)- and anti- Hepatitis B core antibody (HBc)+ (i.e., those who have cleared HBV after infection),
    * Are HBsAg+ with chronic HBV infection (lasting 6 months or longer) and meet conditions below:

      * HBV DNA viral load <100 IU/mL,
      * Have normal transaminase values, or, if liver metastases are present, abnormal transaminases, with a result of AST/ALT <3 × ULN, which are not attributable to HBV infection,
      * Start or maintain antiviral treatment if clinically indicated as per the investigator,
23. Any (attenuated) live vaccine use within 28 days (4 weeks) prior to randomization, while in the study; live vaccines include, but are not limited to, the following: yellow fever, varicella, shingles, measles, mumps, rubella, tuberculosis, rotavirus, influenza,
24. Ongoing or concomitant use of the antiviral drug sorivudine or its chemically related analogs, such as brivudine,
25. Dihydropyrimidine dehydrogenase deficiency (DPD; uracilemia dosage >16 ng/ml), Uracilemia dosing results must be available before inclusion,
26. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of the patient's safety or study results,
27. Known peripheral sensory neuropathy with functional impairment according exclusion criteria n°9) prior to first treatment, according to the Summary of product characteristics (SmPC) of oxaliplatin,
28. Known potentially serious infection, according to the SmPC of 5-FU
29. Has clinically significant active heart disease or myocardial infarction within 6 months given the cardiotoxicity of 5-FU, according to the SmPC of 5-FU,
30. Known history of hypersensitivity to 5-FU, oxaliplatin, or leucovorin, or to any of their excipients, according to the SmPCs of these products.

    Exclusion criteria related to geographical, social, and legal issues
31. Impossibility of submitting to the medical follow-up of the study for geographical, social, or psychiatric illness,
32. Patient under a legal protection regime (guardianship, curatorship, judicial safeguard) or administrative decision or incapable of giving his/her consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) at 4 months | At 4 months
  ORR measured at 4 months post randomization in patients with PD-L1 CPS ≥5 advanced gastric cancer treated by first-line EXL01 plus nivolumab and FOLFOX. ORR at 4 months is defined as the number of patients with a CR or PR evaluated by RECIST v 1.1 criteria divided by the number of patients evaluable.

SECONDARY OUTCOMES:
Overall survival (OS) | Maximum 3 years after randomization
  OS with nivolumab plus FOLFOX with or without EXL01. OS is defined as the time between the date of randomization and the date of death from any cause.
Progression-free survival (PFS) | Maximum 3 years after randomization
  PFS per RECIST v 1.1 and iRECIST of nivolumab plus FOLFOX with or without EXL01.
  PFS is defined as the time from randomization to the date of the first documented PD determined by the Investigator assessment by RECIST 1.1 or death due to any cause, whichever occurs first.
Assessment of safety profile | Maximum 3 years after randomization
  Safety of nivolumab plus FOLFOX with or without EXL01. Safety will be measured by the incidence of Adverse Events (AEs), Serious AEs (SAEs), deaths, laboratory abnormalities, and specific immune-related AEs (hepatitis, colitis, myositis, endocrinopathies).
Duration of response (DoR) | Maximum 3 years after randomization
  DoR with FOLFOX plus nivolumab with or without EXL01. DoR is defined as the time between the date of first documented response (complete response [CR] or partial response [PR]) to the date of the first disease progression, per RECIST 1.1 or death due to any cause, whichever occurs first. For patients who neither progress nor die, the duration of objective response will be censored at the same time they were censored for the primary definition of PFS.
Objective response rate (ORR) | Maximum 3 years after randomization
  ORR per RECIST v 1.1 criteria nivolumab plus FOLFOX with or without EXL01. ORR is defined as the number of patients with the best overall response (BOR) of CR or PR divided by the number of measurable patients with target lesion at baseline. BOR is defined as the best response designation, recorded between the date of randomization and the date of objectively documented progression (per RECIST 1.1) or the date of subsequent anti-cancer therapy, whichever occurs first.
2-year and 3-year OS | At 2 years and 3 years
  2-year and 3-year OS rate of nivolumab plus FOLFOX with or without EXL01
1-year and 2-year PFS | At 1 year and at 2 years
  1-year and 2-year PFS rates per RECIST v 1.1 and iRECIST (immune RECIST) criteria with nivolumab plus FOLFOX with or without EXL01

CONTACTS AND LOCATIONS:
Overall Officials: Romain Cohen, MD, Principal Investigator — Saint-Antoine Hospital
Locations (37):
- France (37):
  - Institut de Cancerologie de L'Ouest Paul Papin, Angers
  - Clinique Sainte Catherine, Avignon
  - Centre Hospitalier Universitaire Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Universitaire Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier Universitaire Clermont Ferrand - Site Estaing, Clermont-Ferrand
  - Centre Hospitalier Henri Mondor, Créteil
  - Centre Georges Francois Leclerc, Dijon
  - Centre Hospitalier Universitaire Grenoble Alpes - Site Nord - Hopital Michallon, La Tronche
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hopital Leon Berard, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Hopital La Timone, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Universitaire Nantes - Hopital Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Cochin, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Saint-Louis, Paris
  - Institut Curie, Paris
  - Institut Gustave Roussy, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Universitaire de Poitiers - Hopital de La Miletrie, Poitiers
  - Centre Hospitalier Universitaire Reims Hopital Robert Debre, Reims
  - Institut Jean Godinot, Reims
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Hopital D'Instruction Des Armées Bégin, Saint-Mandé
  - Centre Hospitalier Saint-Malo, St-Malo
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Centre Hospitalier Universitaire Tours - Hopital Trousseau, Tours
  - CENTRE HOSPITALIER REGIONAL UNIVERSITAIRE DE NANCY Site Brabois, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
  - Medipole Hopital Mutualiste Lyon-Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No